CLINICAL TRIAL: NCT07124039
Title: FIRST-2.0 China: Finerenone FIRST (Finerenone Research of Early Safety and Effectiveness), Part 2.0 in China
Brief Title: An Observational Study Called FIRST-2.0 China to Learn More About the Use of the Study Treatment Finerenone Including How Safe it is and How Well it Works Under Real-world Conditions in a Chinese Population.
Acronym: FIRST-2_CN
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 23030
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — finerenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Finerenone users: Patients with chronic kidney disease and type 2 diabetes mellitus from China who initiate finerenone treatment.
  Interventions: Drug: Finerenone (Kerendia, BAY948862)

INTERVENTIONS:
Drug: Finerenone (Kerendia, BAY948862) — Retrospective cohort analysis using the EHR data from the Tianjin Healthcare and Medical Big Data Platform (China) database.

SUMMARY:
This is a post-authorization safety study (PASS) to describe the real-world use of finerenone in patients with chronic kidney disease (CKD) and type 2 diabetes mellitus (T2D) in China. The study will examine baseline characteristics, comorbidities, and comedications of patients who initiate finerenone treatment. It will also evaluate changes in kidney function markers including estimated glomerular filtration rate (eGFR), urinary albumin-to-creatinine ratio (UACR), and serum potassium levels over time.

The study will assess hyperkalemia incidence, hospitalization rates associated with hyperkalemia, and finerenone dose titration patterns. This retrospective observational cohort study uses data from the Tianjin Healthcare and Medical Big Data Platform covering approximately 15 million residents.

The study aims to provide evidence on finerenone safety and effectiveness in routine clinical practice in China, complementing data from controlled clinical trials. Results will inform healthcare providers about real-world finerenone use patterns and outcomes in Chinese patients with diabetic kidney disease.

ELIGIBILITY:
Inclusion criteria

* Minimum of 12 months continuous enrolment before the index date in the database with medical and pharmacy coverage measured as continuously receiving medical care from health providers contributing to the electronic health record system
* No recorded prescription of finerenone prior to the index date
* Age 18 years or older as of the index date
* Diabetic kidney disease diagnosis by diagnosis texts at any point before (and including) the index date, OR
* T2D diagnosis at any point before (and including) the index date using the same algorithms as in previous studies of the FIRST program, AND

  * CKD stages 2-4 related to eligibility will be defined according to the presence of the following criteria at any point before (and including) the index date:
  * A diagnosis code/text indicating CKD stage 2, 3, 4, or stage unspecified OR
* Two UACR test results ≥30 mg/g separated by at least 90 days and no more than 548 days.

OR

• Two different eGFR test results ≥15 mL/min/1.73 m2 AND <60 mL/min/1.73 m2 separated by at least 90 days and no more than 548 days.

Exclusion criteria

* Type 1 diabetes mellitus identified by diagnosis codes/texts in the patient record on or before the index date
* Kidney cancer identified by diagnosis codes/texts on or before the index date
* Kidney failure on or before the index date, defined as:

  * Two different eGFR test results <15 mL/min/1.73 m2 separated by at least 90 days and no more than 548 days OR
  * Dependence on dialysis (at least 3 sessions over at least 90 days during the baseline period) OR
  * A diagnosis code/text indicating kidney failure or CKD stage 5 OR
  * A recorded diagnosis indicating kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic kidney disease and type 2 diabetes mellitus who initiate finerenone treatment in China
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Descriptive summary of characteristics of patients who initiate finerenone and have CKD and T2D in China. | Up to 365 days
Descriptive summary of comorbidities of patients who initiate finerenone and have CKD and T2D in China. | Up to 365 days
Descriptive summary of comedications of patients who initiate finerenone and have CKD and T2D in China. | Up to 180 days

SECONDARY OUTCOMES:
To describe the routine monitoring of UACR, eGFR, and serum potassium before and after initiating finerenone in patients with CKD and T2D | Up to 32 months
To describe the absolute levels and relative changes over time of UACR, eGFR, and serum potassium after initiating finerenone in patients with CKD and T2D | Up to 32 months
To describe the incidence of hyperkalemia and the incidence of hospitalization associated with a hyperkalemia event after initiating finerenone in patients with CKD and T2D | Up to 32 months
To describe the number of patients who initiate finerenone using a 10 mg dose and the proportion of patients who have up-titrated to a 20 mg dose by 1, 3, 6, and 12 months, respectively, depending on data availability | Up to 32 months

OTHER OUTCOMES:
To describe the baseline characteristics, comorbidities, and comedications | Up to 32 months
  In patients with CKD and T2D in sub-cohorts of patients stratified by baseline UACR level (<30 mg/g, 30-300 mg/g, >300 mg/g), depending on data availability
To describe the absolute levels and relative change over time of UACR, eGFR, and serum potassium after initiating finerenone | Up to 32 months
  In patients with CKD and T2D in sub-cohorts of patients stratified by baseline UACR level (<30 mg/g, 30-300 mg/g, >300 mg/g), depending on data availability
To describe the baseline characteristics, comorbidities, comedications, and the absolute levels and relative change over time of UACR, eGFR, and serum potassium after initiating finerenone | Up to 32 months
  In patients with CKD and T2D in sub-cohorts of patients stratified by baseline UACR and eGFR level (e.g., UACR ≥30 mg/g with eGFR <60 mL/min/1.73m2, UACR ≥30 mg/g with eGFR ≥60 mL/min/1.73m2, UACR <30 mg/g with eGFR <60 mL/min/1.73m2), depending on data availability
To describe the finerenone utilization patterns | Up to 32 months
  In patients with CKD and T2D who initiate finerenone, depending on data availability. Frequency of finerenone use during follow-up, dosing regimen, treatment discontinuation, treatment duration, and treatment persistence will be assessed based on data availability

CONTACTS AND LOCATIONS:
Locations (1):
- Inspur Tianjin Regional Electronic Health Records Database, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
Currently, there is no established plan for the sharing of Individual Patient Data (IPD) from this study. The availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA 'Principles for responsible clinical trial data sharing.' This pertains to the scope, timepoint, and process of data access.
  As such, Bayer commits to considering requests from qualified researchers for patient- / study-level clinical trial data, and documents from clinical trials involving medicines and indications approved in the US and EU. However, this commitment does not reflect an active IPD sharing plan. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Researchers can use www.vivli.org to request access to IPD and documents from clinical studies to conduct research. Information on Bayer's criteria for listing studies is provided in the member section of the portal.